CLINICAL TRIAL: NCT04360226
Title: Assessing the Utility of Peak Inspiratory Flow as a Predictor for COPD Exacerbations
Status: Completed | Type: Observational
Sponsor: Respiratory Effectiveness Group (Other)
Collaborators: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Other Study IDs: REG-RES1801
Record Dates: First submitted 2020-04-19; First posted 2020-04-24 (Actual); Last update posted 2024-04-10 (Actual); Status verified 2024-01

CONDITIONS: Chronic Obstructive Pulmonary Disease
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Non-interventional — Non-interventional, subjects will only have routine testing (blood biomarkers, spirometry, peak inspiratory flow measurements) and be asked to complete questionnaires.

SUMMARY:
This is an international, mulitcentre, observational, prospective study into Peak Inspiratory Flow in COPD patients that aims to: A) Determine the prevalence of suboptimal Peak Inspiratory Flow (PIF) and inadequate inhaler choice and assess the baseline characteristics of these groups. B) Assess the clinical role of PIF and inhaler choice in predicting COPD exacerbations and symptom burden. C) Assess the variability and correlation of PIF with other lung function measurements and CAT score in stable COPD. It is a 12 month study comprising one baseline assessment and 2 follow-up visits at 6 and 12 months.

ELIGIBILITY:
Inclusion Criteria:

1. Spirometry-defined COPD (i.e. post-bronchodilator FEV1/FVC<0.7)
2. Age ≥40 years
3. Smokers or ex-smokers of at least 10 pack-years
4. Clinically stable COPD (no exacerbations in the last 4 weeks)
5. Capable of performing serial lung function tests
6. Prescribed inhaled medication for at least 6 months

Exclusion Criteria:

1. Occurrence of an COPD exacerbation during the previous 4 weeks
2. Have any concomitant chronic respiratory condition other than asthma or bronchiectasis (e.g. cystic fibrosis, lung fibrosis, tuberculosis)
3. Are unable to understand the instructions of the study or to fill the questionnaires
4. Are unwilling to sign the informed consent
5. Are participating in a clinical trial

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: COPD patients, who are clinically stable (4 exacerbations in previous 4 weeks) and have been taking inhaled medications for at least 6 months, but have no other chronic respiratory conditions, other than asthma or bronchiectasis.
Sampling Method: Non-Probability Sample
Enrollment: 400 (Actual)
Dates: Start 2020-12-14 (Actual); Primary Completion 2023-08-01 (Actual); Study Completion 2024-01-25 (Actual)

PRIMARY OUTCOMES:
Prevalence of suboptimal PIF and inadequate inhaler choice. | Baseline
  Determine the prevalence of suboptimal PIF and inadequate inhaler choice.
Exacerbations | 12 months
  Time to first exacerbation associated with different levels of PIF.

SECONDARY OUTCOMES:
PIF and symptom burden | Baseline, 6 and 12 months
  PIF measurements will be correlated with COPD Assessment Test (CAT) Scores. CAT scores range from 0-40 depending on the severity of a persons symptoms; higher scores denote a more severe impact of COPD on a patient's life.
Mortality | 6 and 12 months
  Annual mortality rate associated with different PIF levels.
Variability and correlation of PIF | Baseline, 6 and 12 months
  Variability of PIF over time and the correlation between PIF and other lung function measures (including FEV1, FVC, Inspiratory capacity), CAT scores, T2 markers (nasal polyps and dermatitis) and where available blood biomarkers.
Exacerbation rate | 6 and 12 months
  Annual rate of exacerbations associated with different PIF levels

CONTACTS AND LOCATIONS:
Overall Officials: Omar Usmani, MD, Principal Investigator — National Heart and Lung Institute, Imperial College London & Royal Brompton Hosp
Locations (13):
- University Hospital Sassari, Sassari, Italy
- Mater Dei Hospital, Valletta, Malta
- Singapore (2):
  - Changi General Hospital, Singapore
  - Singapore General Hospital, Singapore
- Ljubljana University Medical Centre, Ljubljana, Slovenia
- South Korea (3):
  - Hanyang University Guri Hospital, Hanyang
  - Seoul St. Mary's Hospital, Seoul
  - Ulsan University Hospital, Ulsan
- Spain (5):
  - Hospital University de Torrecárdenas, Almería
  - University Hospital Vall d'Hebron, Barcelona
  - Hospital Inmaculada HLA, Granada
  - HU Virgen de las Nieves, Granada
  - Hospital Universitario de La Ribera, Valencia

IPD SHARING:
Plan to Share IPD: No